CLINICAL TRIAL: NCT04342286
Title: To Establish a Reproducible Organoid Culture Model With Human Kidney Cancer
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chi Fai NG, Professor, Chinese University of Hong Kong
Other Study IDs: CRE-2019.211
Record Dates: First submitted 2020-04-08; First posted 2020-04-13 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Kidney Cancer
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and Urine sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: Organoid culture — Organoid culture

SUMMARY:
Kidney cancer is one of the ten most common malignancies, and the incidence is increasing in recent year. From Hong Kong Cancer Registry, there was about 670 new cases diagnosed in 2016, and had been increased by 46% compared to 2007.Within the broad classification of kidney cancers, renal cell carcinoma (RCC) accounts for approximately 85% of all cases and greater than 90% of all renal malignancies. Despite the improved understanding and also diagnosis for kidney cancer, still about one fourth of patients will presented at metastatic stage or developed recurrence after initial treatment and required further systemic therapy. Facing the wide range of available options for systemic therapy, the current challenge is how to select the most effective treatment. Unfortunately, there is no good biomarkers available to aid treatment selection.

Currently, there are some approaches to try to test the response of kidney cancer to different chemotherapeutic agents. Previous studies showed that 3D organoid culture model can improve our ability to model tumor behavior. Organoid culture technology may provide opportunities for new drug development and drug screening.

In this study, investigators aim to establish a reliable and effective method to cultivate kidney cancer cells, then will provide researchers for further information on personalized and targeted therapy on kidney cancer for local Hong Kong patients.

DETAILED DESCRIPTION:
Kidney cancer is one of the ten most common malignancies, and the incidence is increasing in recent year. From Hong Kong Cancer Registry, there was about 670 new cases diagnosed in 2016, and had been increased by 46% compared to 2007. The rapid increase in incidence is partly due to the greater prevalence of putative risk factors including smoking, obesity, and hypertension, as well as improvements in diagnostic imaging. Within the broad classification of kidney cancers, renal cell carcinoma (RCC) accounts for approximately 85% of all cases and greater than 90% of all renal malignancies.

Despite the improved understanding and also diagnosis for kidney cancer, still about one fourth of patients will presented at metastatic stage or developed recurrence after initial treatment and required further systemic therapy. Fortunately, with recent advances in the development of novel therapeutic agents, there are many potential effective treatments available for patients, including tyrosine kinase inhibitors, mammalian target of rapamycin (mTOR) inhibitors, immune checkpoint blockers etc. Facing the wide range of available options for systemic therapy, the current challenge is how to select the most effective treatment for individual patients, in particular as the first line therapy.

Currently, there are some guidelines, basing on the clinical parameters and tumor subtype and grading, for selection of therapy for patients.Unfortunately, there is no good biomarkers available to aid treatment selection. As there is increasing recognition of inter-tumor variation, therefore, there is a need to develop more personalized approach to assess the treatment response of individual patient / cancer to the panel of available drugs, in order to select the best options for each patient.

Three-dimensional (3D) organoid culture model and its potential advantages Organoid technology has recently emerged to become an independent research tool and can provide opportunities for new drug development and drug screening. Organoids are cell-derived in vitro 3D organ constructs which allow the study of many biological processes. This specific model can be developed from embryonic stem cells (ESCs), induced pluripotent stem cells (iPSCs), somatic SCs, and cancer cells in specific 3D culture systems. These groundbreaking 3D tissues were first created in the laboratory in small scale and closely resembled the parent organ in vivo in terms of its structure and function. The major benefits of the 3D organoid culture model include, firstly, it contains multiple cell types comparable with the in vivo counterpart; secondly, the cells inside the 3D structure can organize similarly to the primary tissue; and lastly, it functions specifically like the parent organ. With the scaffold supporting and the nascent phenotype needed, emerging 3D culture methods can improve our ability to model tumor behavior in vitro and provide a native environment for different research purposes, such as cell behavior, tissue repair, drugs screening and mutation monitoring. Development of kidney cancer organoid Different studies have demonstrated that gastrointestinal cancers organoid models provide better prediction to a patient's treatment responses. There is limited publication on successful 3D kidney cancer organoid recently, and the one published by Batchelder CA in 2015 had analyzed limited amount of genes. Besides, majority of the cases reported had been undergone 2D culture on plasticwares before implanting inside the 3D scaffold, which may offer the chance of cells selection.Lacking a widely acceptable 3D kidney cancer model, this pushes the need to develop a reproducible kidney cancer organoid system for better drug selection on significant heterogeneity cancers. In our study, total cells will be mixed with the Matrigel scaffold without any manipulation or culture selection, and more advance Next Generation Sequencing will be used to evaluate the genetic similarity of the culture organoids and the primary tissues. Starting as a major technological breakthrough, 3D organoids are now more firmly established as an essential tool in biological research and have important implications for clinical use. In the future, successful expansion of the model can provide a platform to identify the most effective personalized treatment option and improve the treatment outcome of kidney cancer patients.

Therefore, investigator proposed to establish a sustainable human kidney tumor 3D Matrigel culture system with a stable phenotype from local population. Investigators hypothesize that the successful of our project would produce reliable and effective method to cultivate kidney cancer cells from our local patients, and will provide personalized and targeted therapy on kidney cancer for local Hong Kong patients.

ELIGIBILITY:
Inclusion Criteria:

* Male patients > 18 years old
* Patients suffered from renal cell carcinoma require surgical removal of kidney

Exclusion Criteria:

* Patients fail to provide informed consent
* The collection of tissue will affect the pathological interpretation of the specimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a methodology development project aiming at developing a reproducible 3D kidney cancer organoid model. Twenty patients suffered from renal cell carcinoma and planned for surgical treatment will be recruited for this study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-02-22 (Actual); Study Completion 2021-02-22 (Actual)

PRIMARY OUTCOMES:
To establish a sustainable human kidney tumor 3D Matrigel culture system with a stable phenotype | 2 years
  A Cell culture is successful when organoids grow from dividing cells

SECONDARY OUTCOMES:
The identicality of histopathological detail and genomic information of the kidney cancer organoid compared with the original primary tissue | 2 years
  The identicality is assessed by the histopathological detail and the genomic information of the kidney cancer organoid compared with the original primary tissue
The tumorigenicity ability of the kidney cancer organoid in nude mice | 2 years
  The tumorigenicity ability will be assessed by nude mice injection

CONTACTS AND LOCATIONS:
Overall Officials: Chi Fai NG, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mer AS, Ba-Alawi W, Smirnov P, Wang YX, Brew B, Ortmann J, Tsao MS, Cescon DW, Goldenberg A, Haibe-Kains B. Integrative Pharmacogenomics Analysis of Patient-Derived Xenografts. Cancer Res. 2019 Sep 1;79(17):4539-4550. doi: 10.1158/0008-5472.CAN-19-0349. Epub 2019 May 29. PMID 31142512
- [Background] Batchelder CA, Martinez ML, Duru N, Meyers FJ, Tarantal AF. Three Dimensional Culture of Human Renal Cell Carcinoma Organoids. PLoS One. 2015 Aug 28;10(8):e0136758. doi: 10.1371/journal.pone.0136758. eCollection 2015. PMID 26317980
- [Background] Alley MC, Scudiero DA, Monks A, Hursey ML, Czerwinski MJ, Fine DL, Abbott BJ, Mayo JG, Shoemaker RH, Boyd MR. Feasibility of drug screening with panels of human tumor cell lines using a microculture tetrazolium assay. Cancer Res. 1988 Feb 1;48(3):589-601. PMID 3335022
- [Background] Drost J, Karthaus WR, Gao D, Driehuis E, Sawyers CL, Chen Y, Clevers H. Organoid culture systems for prostate epithelial and cancer tissue. Nat Protoc. 2016 Feb;11(2):347-58. doi: 10.1038/nprot.2016.006. Epub 2016 Jan 21. PMID 26797458
- [Background] Gao H, Korn JM, Ferretti S, Monahan JE, Wang Y, Singh M, Zhang C, Schnell C, Yang G, Zhang Y, Balbin OA, Barbe S, Cai H, Casey F, Chatterjee S, Chiang DY, Chuai S, Cogan SM, Collins SD, Dammassa E, Ebel N, Embry M, Green J, Kauffmann A, Kowal C, Leary RJ, Lehar J, Liang Y, Loo A, Lorenzana E, Robert McDonald E 3rd, McLaughlin ME, Merkin J, Meyer R, Naylor TL, Patawaran M, Reddy A, Roelli C, Ruddy DA, Salangsang F, Santacroce F, Singh AP, Tang Y, Tinetto W, Tobler S, Velazquez R, Venkatesan K, Von Arx F, Wang HQ, Wang Z, Wiesmann M, Wyss D, Xu F, Bitter H, Atadja P, Lees E, Hofmann F, Li E, Keen N, Cozens R, Jensen MR, Pryer NK, Williams JA, Sellers WR. High-throughput screening using patient-derived tumor xenografts to predict clinical trial drug response. Nat Med. 2015 Nov;21(11):1318-25. doi: 10.1038/nm.3954. Epub 2015 Oct 19. PMID 26479923
- [Background] Huch M, Gehart H, van Boxtel R, Hamer K, Blokzijl F, Verstegen MM, Ellis E, van Wenum M, Fuchs SA, de Ligt J, van de Wetering M, Sasaki N, Boers SJ, Kemperman H, de Jonge J, Ijzermans JN, Nieuwenhuis EE, Hoekstra R, Strom S, Vries RR, van der Laan LJ, Cuppen E, Clevers H. Long-term culture of genome-stable bipotent stem cells from adult human liver. Cell. 2015 Jan 15;160(1-2):299-312. doi: 10.1016/j.cell.2014.11.050. Epub 2014 Dec 18. PMID 25533785
- [Background] Li M, Izpisua Belmonte JC. Organoids - Preclinical Models of Human Disease. N Engl J Med. 2019 Feb 7;380(6):569-579. doi: 10.1056/NEJMra1806175. No abstract available. PMID 30726695
- [Background] Li YY, Chung GT, Lui VW, To KF, Ma BB, Chow C, Woo JK, Yip KY, Seo J, Hui EP, Mak MK, Rusan M, Chau NG, Or YY, Law MH, Law PP, Liu ZW, Ngan HL, Hau PM, Verhoeft KR, Poon PH, Yoo SK, Shin JY, Lee SD, Lun SW, Jia L, Chan AW, Chan JY, Lai PB, Fung CY, Hung ST, Wang L, Chang AM, Chiosea SI, Hedberg ML, Tsao SW, van Hasselt AC, Chan AT, Grandis JR, Hammerman PS, Lo KW. Exome and genome sequencing of nasopharynx cancer identifies NF-kappaB pathway activating mutations. Nat Commun. 2017 Jan 18;8:14121. doi: 10.1038/ncomms14121. PMID 28098136
- [Background] McKay RR, Bosse D, Choueiri TK. Evolving Systemic Treatment Landscape for Patients With Advanced Renal Cell Carcinoma. J Clin Oncol. 2018 Oct 29:JCO2018790253. doi: 10.1200/JCO.2018.79.0253. Online ahead of print. PMID 30372392
- [Background] Meijer TG, Naipal KA, Jager A, van Gent DC. Ex vivo tumor culture systems for functional drug testing and therapy response prediction. Future Sci OA. 2017 Mar 27;3(2):FSO190. doi: 10.4155/fsoa-2017-0003. eCollection 2017 Jun. PMID 28670477
- [Background] Morizane R, Bonventre JV. Kidney Organoids: A Translational Journey. Trends Mol Med. 2017 Mar;23(3):246-263. doi: 10.1016/j.molmed.2017.01.001. Epub 2017 Feb 7. PMID 28188103
- [Background] van de Wetering M, Francies HE, Francis JM, Bounova G, Iorio F, Pronk A, van Houdt W, van Gorp J, Taylor-Weiner A, Kester L, McLaren-Douglas A, Blokker J, Jaksani S, Bartfeld S, Volckman R, van Sluis P, Li VS, Seepo S, Sekhar Pedamallu C, Cibulskis K, Carter SL, McKenna A, Lawrence MS, Lichtenstein L, Stewart C, Koster J, Versteeg R, van Oudenaarden A, Saez-Rodriguez J, Vries RG, Getz G, Wessels L, Stratton MR, McDermott U, Meyerson M, Garnett MJ, Clevers H. Prospective derivation of a living organoid biobank of colorectal cancer patients. Cell. 2015 May 7;161(4):933-45. doi: 10.1016/j.cell.2015.03.053. PMID 25957691
- [Background] Williams JA. Using PDX for Preclinical Cancer Drug Discovery: The Evolving Field. J Clin Med. 2018 Mar 2;7(3):41. doi: 10.3390/jcm7030041. PMID 29498669
- [Background] Xu H, Lyu X, Yi M, Zhao W, Song Y, Wu K. Organoid technology and applications in cancer research. J Hematol Oncol. 2018 Sep 15;11(1):116. doi: 10.1186/s13045-018-0662-9. PMID 30219074
- See also: Hong Kong Cancer Registry — http://www3.ha.org.hk/cancereg/allagesresult.asp